CLINICAL TRIAL: NCT00163917
Title: Predicting the Effectiveness of Virtual Reality Relaxation on Pain and Anxiety When Added to PCA Morphine in a Population of Burn Patients Having Dressing Changes
Brief Title: A Study of the Effectiveness of Virtual Reality Relaxation Combined With Patient-Controlled Analgesia (PCA) Morphine for Those Undergoing Burn Dressing Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 107/ 04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2005-09

CONDITIONS: Anxiety; Pain
Keywords: Hypnosis; Analgesia
MeSH Terms: conditions — Anxiety Disorders; Pain; Agnosia

INTERVENTIONS:
Device: Virtual reality relaxation

SUMMARY:
The purpose of this study is to evaluate whether a sub-population of patients with burn injuries needing dressing changes respond to virtual reality (VR) utilising relaxation themes with improved pain and anxiety scores, when added to PCA morphine and background analgesic therapy.

DETAILED DESCRIPTION:
Pain associated with burn dressing changes does not arise purely from a physical source; it is also commonly influenced by psychological factors. The anticipation that accompanies a dressing change has the potential to set up fear and heightened anxiety as the patient is aware that at a predetermined time other people will manipulate injured areas on his/her body.

Many techniques of analgesia have been advocated in burn dressing changes. Opiates have been the mainstay, and many techniques for their administration have been described. In particular the use of background plus PCA administration of opiates has been demonstrated to be superior to PCA administration alone. Another analgesic/dissociative agent commonly described for these procedures is Ketamine. Both opiates and ketamine have limitations in that they cause unfavourable side effects such as respiratory depression, sedation and nausea and vomiting in the case of opiates and respiratory depression, hallucinations and unpleasant dreams in the case of ketamine. Other problems relating to the use of opiates and ketamine relate to the approach of treating a multifaceted experience such as burn dressing pain solely with pharmacotherapy.

The need for psychological interventions in burn dressings has been highlighted by many researchers. In particular, Ptacek noted that burn patients experiencing more anxiety tended to have higher ratings of pain, while those with larger areas of burns reported more affective pain and greater variability in pain ratings.

There is strong consistency among reviewers for recommending the addition of adjunctive therapies of a psychological nature for managing patients having burn dressing changes. Patterson et.al in particular is of the belief that burn patients having dressing changes are more amenable to hypnotherapy as an analgesic adjunct.

The nature of psychological interventions examined by researchers have included hypnosis (where strong suggestions were aimed at reducing tension, anxiety, and sensation of pain), rapid induction analgesia, simple stress reducing strategies, attention and information, and autohypnosis. While some have conducted prospective trials which involve large numbers of patients, only one trial actually made mention of randomizing participants. Most other reports examining psychological therapies have been at the case report level.

While most of these trials and case reports have reported favourable outcomes, no single trial has been able to consistently show a significant reduction of pain scores and anxiety ratings and analgesic consumption.

Virtual Reality (VR) assisted techniques that modify psychological well-being are beginning to play a role in clinical practise and in research. There are currently two publications, one a case report and another a prospective randomized trial which specifically examine the role of VR in the context of painful procedures associated with burn injuries. The randomized crossover trial by Hoffman et.al in 6 patients having physical therapy utilising immersive VR found a significant reduction in pain ratings in all patients, while Patterson et.al described the successful use of VR hypnosis in one "difficult" patient which had lasting effects for up to 48 hours.

Reviews of psychological therapies for patients having burn dressing changes have addressed the need for more systematic controlled trials to supplement existing evidence and more clearly define the role of such interventions. Coupled with this is the need for more knowledge as to the most appropriate psychological intervention and the ideal situations where it will prove most beneficial. Patterson feels that there is good anecdotal evidence that burn patients have a particular propensity to respond to adjunctive therapies incorporating hypnosis. Hypnosis screening among burn patients involving the hypnotic induction profile demonstrated a link between high hypnotizability and the experience of more intense arousal, greater avoidance and more significant feelings of intrusiveness.

We propose to conduct a prospective randomized trial which looks at the effect that VR relaxation has when combined with PCA morphine in a group of patients having potentially painful dressing changes. In addition we want to isolate patients who have high susceptability to hypnosis and compare their ratings of pain, anxiety and opiate requirement with patients of lesser susceptibility. Our hypothesis is that patients with higher susceptibility to hypnosis stand to gain most from the addition of VR to their pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury
* Scheduled for painful dressing changes
* Conscious
* Comprehension of PCA and virtual reality device
* Comprehension of the English language

Exclusion Criteria:

* Patient refusal
* Psychotic disease
* Paranoid disease
* Unstable dissociative disorder
* Borderline personality disorder
* Phobias relevant to water/drowning
* Epilepsy/propensity to fitting
* Morphine allergy
* Acute brain syndrome
* Chronic brain syndrome
* Physically unable to administer PCA
* Severe burns involving the head
* Visual impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-09

PRIMARY OUTCOMES:
Association between hypnotic susceptibility and pain scores
Association between hypnotic susceptibility and anxiety scores

SECONDARY OUTCOMES:
Measurement of pain by visual analogue scale (VAS)
Measurement of anxiety by Burns Specific Anxiety Rating by VAS
Rating of hypnotic susceptibility and morphine use
Satisfaction rating
Morphine use
Incidence of side effects relating to morphine and VR

CONTACTS AND LOCATIONS:
Overall Officials: Alex Konstantatos, MBBS, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia